CLINICAL TRIAL: NCT04752280
Title: Glioblastoma Radiotherapy Using IMRT or Proton Beams
Acronym: GRIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRIPS
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Proton irradiation (Experimental): Irradiation applied with protons
  Interventions: Radiation: Proton irradiation
- Arm B: Photon IMRT (Active Comparator): Photon irradiation applied as intensity-modulated radiotherapy
  Interventions: Radiation: Photon irradiation

INTERVENTIONS:
Radiation: Proton irradiation — proton irradiation applied as follows: 30 x 2 Gy(RBE) 33 x 1,8 Gy (RBE), or 15 x 2,67 Gy (RBE)
  Arms: Arm A: Proton irradiation
Radiation: Photon irradiation — proton irradiation applied as follows: 30 x 2 Gy 33 x 1,8 Gy, or 15 x 2,67 Gy
  Arms: Arm B: Photon IMRT

SUMMARY:
Radiation therapy is an integral part of the multimodal primary therapy of glioblastomas. As the overall prognosis in this tumor entity remains unfavorable, current research is focused on additional drug therapies, which are often accompanied by increases in toxicity. By using proton beams instead of photon beams, it is possible to protect large parts of the brain which are not affected by the tumor more effectively. An initial retrospective matched-pair analysis showed that this theoretical physical benefit is also clinically associated with a reduction in toxicity during therapy and in the first few months thereafter. The aim of the GRIPS study is to prospectively test this clinical benefit in a randomized, open-label Phase III study. Patients are treated in the study using either modern photon radiation techniques (standard arm) or proton beams (experimental arm). The primary endpoint is the cumulative toxicity CTC grade 2 and higher in the first 4 months. Secondary endpoints include overall survival, progression-free survival, quality of life, and neurocognition.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed gliomblastoma WHO IV (operated or after biopsy)
* Indication for radiotherapy / radiochemotherapy
* Informed consent
* KI ≥ 60% or ECOG 0/1
* Age ≥ 18 years
* Sufficient effective contraception

Exclusion Criteria:

* Patient is not able to consent
* Previous radiotherapy in the brain or skull base
* Active medical implants for which there is no ion radiation authorization at the time of treatment (e.g., cardiac pacemaker, defibrillator, ...)
* Contraindication to MRI imaging
* Simultaneous participation in another clinical trial that could influence the outcome of this study or other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2027-10-19 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of toxicity | from start of radiotherapy until progress (max. month 4)
  Cumulative rate of toxicity ≥ grade 2 (until progress (max. month 4))

SECONDARY OUTCOMES:
Progression free survival | 1 year and 2 years
  Progression free survival
Overall survival | 1 year and 2 years
  Overall survival
Acute Toxicity | start of therapy until 6 weeks after end of therapy (end of therapy up to month 4)
  according to CTC AE V5.0
Late Toxicity | 6 weeks after end of therapy (end of therapy up to month 4)
  according to CTC AE V5.0
Quality of life according to EORTC QLQ-C30 | 1 year and 2 years
  according to EORTC QLQ-C30
Quality of life according to EORTC QLQ-BN20 | 1 year and 2 years
  according to EORTC QLQ-BN20
Neurocognition | 1 year and 2 years
  according to Hopkins Verbal Learning Test-Revised
Measuring number of Lymphocytes count | end of therapy up to month 4

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Klinikum Stuttgart, Stuttgart

REFERENCES:
- [Derived] Konig L, Jakel C, von Knebel Doeberitz N, Kieser M, Eberle F, Munter M, Debus J, Herfarth K. Glioblastoma radiotherapy using Intensity modulated Radiotherapy (IMRT) or proton Radiotherapy-GRIPS Trial (Glioblastoma Radiotherapy via IMRT or Proton BeamS): a study protocol for a multicenter, prospective, open-label, randomized, two-arm, phase III study. Radiat Oncol. 2021 Dec 20;16(1):240. doi: 10.1186/s13014-021-01962-8. PMID 34930368